CLINICAL TRIAL: NCT04424303
Title: Evaluation of the Clinical Benefit of ToFAcitinib Treatment in Patients With Moderate to Severe Ulcerative Colitis Under Real-life Conditions of Use: TOFAst Study
Brief Title: Tofacitinib in Adult Patients With Moderate to Severe Ulcerative Colitis
Acronym: TOFAST
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921360; TOFAst study (Other: Alias Study Number)
Record Dates: First submitted 2020-06-08; First posted 2020-06-09 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis, Tofacitinib, France, Real world data
MeSH Terms: conditions — Colitis, Ulcerative | interventions — tofacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients prescribed tofacitinib: Patients with a confirmed diagnosis of moderate to severe ulcerative colitis initiating tofacitinib as per the French summary of product characteristics (SmPC).
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — Observational study

SUMMARY:
This is an observational prospective study with two years of follow-up, designed to evaluate the effectiveness of tofacitinib in patients with moderate to severe ulcerative colitis in French clinical practice

DETAILED DESCRIPTION:
TO FAst is a non-interventional study in France with primary objective to describe the clinical benefit of tofacitinib 1 year after its initiation for the treatment of moderate to severe UC in routine clinical practice. The study will also make it possible to report the clinical benefit 2 years after its initiation, to search for predictors of clinical benefit, improve our understanding of the efficacy of treatment in a real-life setting (in terms of response and speed of response), describe the characteristics of patients starting a treatment by tofacitinib, its real-life patterns of use as well as patient adherence to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 18 years old or above
* Patients with confirmed diagnosis of moderate to severe ulcerative colitis
* Patients for whom gastroenterologist decides to initiate treatment with tofacitinib as per the French SmPC
* Patients informed about the study procedures and receiving an information letter signed by the investigator

Exclusion Criteria:

* Patients who have already received tofacitinib treatment before baseline
* Patients that fulfill any of the contrindications according to the latest version of the SmPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with moderate to severe Ulcerative Colitis initiating tofacitinib treatment as per the French Summary of product characteristics (SmPC)
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with clinical benefit one year after initiation of tofacitinib treatment. | Week 52
  The definition of clinical benefit is independent of the discontinuation or not of tofacitinib treatment during the observation period.
  Clinical benefit at year is defined on the basis of symptomatic remission evaluated with the PRO2 score ≤1 (absence of rectal bleeding and a stool frequency score between 0 and 1)*. Patients who died or who had a colectomy or used another biologic/anti-JAK/immunosuppressant will be considered to be non-responders, as well as patients who used oal corticosteroids for UC, (regardless of the treatment duration) during the 3 months preceding the end of the observation period.
  The clinical benefit of tofacitinib is independent of the administration or not of 5-ASA, or corticosteroids (not complying with the above definition) during the observation period (between 0 and 1 year).

SECONDARY OUTCOMES:
Proportion of patients with clinical benefit of tofacitinib at 2 years | week 104
Predictors of the clinical benefit at one year identified from the available baseline data | Week 52
Proportion of patients in clinical remission and still receiving tofacitinib | Week 52 and Week 104
  Clinical remission is defined as partial Mayo score (PMS) <2
Proportion of patients in clinical remission without corticosteroids (oral or topical with systemic effects for UC) | Week 52 and week 104
Proportion of patients with short-term clinical response for patients still treated with tofacitinib | Approximately week 8 and 16
  Clinical response is defined as a reduction in partial Mayo score ≥ 3 points and ≥ 30% with respect to baseline, with a concomitant reduction in rectal bleeding sub-score ≥ 1 point (absolute sub-score of 0 or 1).
Proportion of patients with biological response during the observation period | Week 52 and 104
  Biological response is defined as 50% reduction in the initial value of CRP or Fecal Calprotectine (FCP)
Proportion of patients with endoscopic improvement during the observation period | Week 52 and 104
  endoscopic improvement is defined as endoscopic subscore of 0 or 1
Proportion of patients in sustained clinical remission | Week 52 and 104
  Clinical remission is defined as partial Mayo score (PMS) <2 at 52 and 104 weeks
Time to loss of response to tofacitinib treatment in patients after dose reduction to 5 mg BID at the end of induction | Week 8, 16, 24, 72, 52 and 104
  The clinical loss of response is defined by a recrudescence of the symptoms that lead to a systemic therapeutic intervention (return to previous dose of tofacitinib or corticosteroid therapy, or an immunosuppressant or biologic/other anti-JAK)
Proportion of patients with extraintestinal manifestations at each visit | Week 8, 16, 24, 72, 52, 104
Proportion of patients with a colectomy during study follow-up and time of occurrence | Week 8, 16, 24, 72,52 and 104
Characteristics of patients and UC, on the basis of all the data collected at baseline | Week 104
Description of the changes in the rectal bleeding and stool frequency subscores during the first 2 weeks after initiation of tofacitinib therapy | 14 days
  (self-assessment by patients)
Change in patient quality-of-life evaluated from the SIBDQ questionnaire between baseline and 1 year, baseline and 2 years, and between 1 and 2 years | Week 52, Week 52 to week 104 and week 104
Change in adherence to tofacitinib treatment during each visit | Week 8, 16, 24, 72, 52, 104
  Using MARS questionnaire
Proportion of patients with serious and non-serious adverse events. | Week 8, 16, 24,72,52 and 104

OTHER OUTCOMES:
Proportion of patients with a clinical response* 1 year and 2 years after initiation of tofacitinib | Week 52 and 104
  Reduction in partial Mayo score ≥ 3 points and ≥ 30% with respect to baseline, with a concomitant reduction in rectal bleeding sub-score ≥ 1 point (absolute sub-score of 0 or 1).

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (38):
- France (38):
  - Clinique de l Europe, Amiens
  - Hopital Sud, Amiens
  - Hopital Jean Minjoz, Besançon
  - Hopital de La Cote de Nacre, Caen
  - Centre Hospitalier de Cahors, Cahors
  - Infirmerie Protestante de Lyon, Caluire-et-Cuire
  - Hopital Trousseau, Chambray-lès-Tours
  - Hopital D'Estaing, Clermont-Ferrand
  - Aphp - Hopital Beaujon, Clichy
  - Ch Intercommunal de Creteil, Créteil
  - Ch Dunkerque, Dunkirk
  - Hopital Albert Michallon, La Tronche
  - Ch Bicetre, Le Kremlin-Bicêtre
  - CH Le Mans, Le Mans
  - Ch Emile Roux, Le Puy-en-Velay
  - Hopital Claude Huriez, Lille
  - Ch Saint Joseph Saint Luc, Lyon
  - Ch Montfermeil, Montfermeil
  - Clinique Beau Soleil, Montpellier
  - Hopital Saint Eloi, Montpellier
  - Chu Nantes, Nantes
  - Clinique Jules Verne, Nantes
  - Hopital de L'Archet, Nice
  - Hopital Caremeau, Nîmes
  - Hopital Europeen Georges Pompidou, Paris
  - Aphp - Hopital Saint Louis, Paris
  - Groupe Hospitalier Saint Joseph, Paris
  - Chu Bichat Claude Bernard, Paris
  - Chu de Bordeaux - Hopital Haut Leveque, Pessac
  - CHU LYON, Pierre-Bénite
  - Ch Annecy Genevois, Pringy
  - Chu Rennes, Rennes
  - Hopital Nord, Saint-Priest-en-Jarez
  - Clinique Pasteur, Toulouse
  - Hopital Rangueil, Toulouse
  - Ch Valence, Valence
  - Ch Valenciennes, Valenciennes
  - Groupe Hospitalier Mutualiste Les Portes du Sud, Vénissieux

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921360